CLINICAL TRIAL: NCT07017595
Title: Improving the Accessibility of Gender-affirming Voice Training With Visual-acoustic Biofeedback
Brief Title: Gender-affirming Voice Training With Visual Feedback
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was terminated by NIH in 2025 with a statement that the research no longer meets agency priorities.
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); New York University (Other); University of Central Florida (Other)
Responsible Party: Principal Investigator, Vesna D Novak, PhD, Associate Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0831; R21DC021537 (NIH)
Record Dates: First submitted 2025-05-24; First posted 2025-06-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Transgender Women; Voice Alteration
Keywords: transgender; gender-affirming voice and communication training; voice training; voice-gender incongruence; transgender women; voice alteration; voice change
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: There will be only one group. Each participant will take part in the same protocol (4 virtual training sessions + "homework" between sessions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experiment group (Experimental): This group will be given access to our prototype software for pitch and resonance training. They will go through 4 virtual sessions of expert-guided voice training, with the software used as part of the sessions, and will use the software on their own between sessions.
  Interventions: Behavioral: Visual-acoustic biofeedback: experimental

INTERVENTIONS:
Behavioral: Visual-acoustic biofeedback: experimental — Visual-acoustic biofeedback treatment incorporates elements of traditional voice training, including auditory models, verbal descriptions of articulator placement, and cues for repetitive motor practice using images and diagrams of the vocal tract as visual aids. Our experimental software will provide several options for visualizing the fundamental frequency of the voice (for targets involving vocal pitch) and for visualizing vocal tract resonances. Custom targets for pitch and resonance will be created for each participant based on their baseline voice characteristics and personal voice goals. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments influence the proximity of their output to the target.

SUMMARY:
The goal of this clinical trial is to learn if prototype software can be used to train vocal pitch and resonance in trans women. The main questions it aims to answer are:

* How regularly would trans women use the prototype voice training software as "homework" between human-led voice training sessions?
* In such a setting, how usable and motivating would the training software be?

Participants will first have their voice measured, then take part in four virtual sessions (one per week) led by a speech-language pathologist. In each session, the clinician will guide the participant through several voice exercises both with and without the software. Participants will be asked to use the software to exercise on their own for about 2x 15 minutes a day between virtual sessions.

DETAILED DESCRIPTION:
In an initial virtual assessment session (conducted via a password-protected Zoom room), a researcher will explain the protocol, obtain informed consent, collect participant demographics and other self-report data, and obtain baseline recordings of the participant's voice while speaking different utterances.

After the initial assessment session, each participant will take part in four virtual training sessions (on day 1, after approximately 1 week, after approximately 2 weeks, after approximately 3 weeks) provided on an individual basis by a certified speech-language pathologist (SLP).

In the first session (1 hour), the SLP will assess each participant's baseline ability to modify their pitch and resonance and will introduce the voice training software. They will provide strategies that participants may use to manipulate their pitch or resonance (e.g., for resonance, changing the positioning of the tongue in their mouth or changing the shape of the lips). For the remainder of the session, the SLP will guide the participant through exercises deemed appropriate to the participant's ability, both with and without the software. At the end of the session, the SLP will prescribe pitch and/or resonance exercises to be performed at home with the voice training software, with a suggested duration of 2x 15 minutes each day. Additional one-hour virtual training sessions with the SLP will be held at the end of weeks 1, 2, and 3.

Between sessions, participants will be asked to exercise on their own and report the duration and type of practice using a self-report log, though there will be no mechanism to enforce the unsupervised exercise.

After the last training session, participants will take part in a final assessment session where the same recordings as in the initial assessment session will be obtained again and additional self-report data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Native speaker of American English - must have been exposed to it by the age of 6.
* Assigned male at birth, currently identifies as transgender.
* Currently interested in gender-affirming voice training.
* Has access to a computer and quiet room for performing voice training.
* Able to pass a pure-tone hearing screening at 20dB HL.

Exclusion Criteria:

* Current or previous diagnosed speech, language or hearing problems (besides voice-gender dysphoria).
* Neurological disorder or disease (e.g., Parkinson's, tremor) or impacted nerve function to the larynx (e.g., paralysis/paresis of the vocal fold).
* Respiratory disease (e.g., asthma).
* Nasopharyngeal pathology or anatomical abnormality.
* Previous voice feminization surgery.
* Engaged in other gender-affirming voice training during period of study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender women and nonbinary transfeminine participants
Enrollment: 6 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Intrinsic Motivation Inventory (IM) | During the first and fourth intervention sessions
  The IMI is a patient-reported outcome measure that collects information about participants' experience of interacting with a particular task or technology. The total instrument consists of 45 items under seven subcategories (Interest/Enjoyment, Perceived Competence, Effort/Importance, Pressure/Tension, Perceived Choice, Value/Usefulness, and Relatedness). We will use an 8-item version of the scale that has been adopted in previous lab-based studies on motivation, including several by our group. The IMI will be administered after participants are first exposed to their assigned software in the first training session, and again at the end of the three-week training period.
Time on task | Data collected throughout the three-week duration of training
  Participants will be provided with a standard log to record their minutes of practice over the three-week training period. The total number of self-reported minutes of practice completed will serve as a primary outcome measure of interest and will be compared to the a priori requested 30 minutes per day.

SECONDARY OUTCOMES:
Acoustically measured change over time | Baseline (pre-intervention) and immediately after the last intervention session
  Participants will be recorded producing a brief speech sample in their "best feminine voice" at the start and end of participation. Mean pitch, pitch range, and mean F2 frequency will be calculated for each sample. Change in these values from pre- to post-training will be used to assess the effects of the brief duration of training provided. This is considered a secondary outcome since the duration of the protocol (3 weeks) is significantly shorter than full gender-affirming voice training regimens and effects on this outcome may not yet be visible.
Self-Efficacy Scale for Voice Modification in Trans Women | Baseline (pre-intervention) and immediately after the last intervention session
  The SES-VMTW is patient-reported outcome measure consisting of 19 items that ask participants to rate their own ability to adjust the characteristics of their voice (e.g., "I can raise the pitch of my voice") and their ability to complete voice exercises under different conditions of practice (e.g., "I can organise a quiet place to practice my voice exercises"). We will administer the full questionnaire at pre- and post-training time points.

OTHER OUTCOMES:
System Usability Scale (SUS) | Immediately after training
  The System Usability Scale is a simple ten-item scale attitude Likert scale giving a global view of subjective assessments of usability. It has a range of 0-100, with higher scores indicating better usability. The scale will be used to collect participants' opinions about the voice training software.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all anonymized data with other researchers. This is expected to include questionnaire answers and acoustic metrics extracted from data, but not, e.g., audio recordings or specific participant data that would allow the participant to be individually identified (e.g., date of birth).